CLINICAL TRIAL: NCT00038597
Title: Phase II Study of SCH66336, A Farnesyltransferase Inhibitor in Chronic Myelogenous Leukemia (CML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM01-072
Record Dates: First submitted 2002-06-03; First posted 2002-06-04 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Myelogenous Leukemia, Chronic
Keywords: Philadelphia chromosome positive CML; Myelogenous Leukemia, Chronic, Chronic Phase; Myelogenous Leukemia, Chronic, Accelerated Phase
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid; Bronchiolitis Obliterans Syndrome | interventions — lonafarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SCH66336

SUMMARY:
The goal of this research is to see if giving the drug SCH66336 by mouth can improve the disease in patients with chronic or accelerated phase CML. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Objectives for this study are two-fold:

1. To determine the efficacy of SCH66336 in patients with chronic phase and accelerated phase CML in relation to response rate, duration of response, and survival.
2. To assess the toxicity of SCH66366 in these patients.

ELIGIBILITY:
* Diagnosis of Philadelphia chromosome (Ph) -positive CML in chronic or accelerated phase;
* Failure to respond to or intolerance to imatinib mesylate (Gleevec);
* Age >/= 16 years;
* Life expectancy of >/= 2 months;
* Performance status 2 or better (Zubrod);
* Adequate renal and hepatic functions (creatinine and bilirubin </= 2 mg/dl);
* Adequate cardiac function;
* Not candidates for or have refused allogeneic transplantation;
* Patients should not be receiving azoles (ketoconazole, itraconazole, fluconazole), macrolides, HIV protease inhibitors, cyclosporin or anti-seizure drugs (phenobarbital, phenytoin, carbamazepine), rifampin or isoniazid.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2001-04-30 (Actual); Primary Completion 2004-05-07 (Actual); Study Completion 2004-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- MDAnderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org